CLINICAL TRIAL: NCT00005471
Title: Anxiety and Cardiovascular Autonomic Control
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4953; R01HL054098 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To evaluate the hypothesis that chronic anxiety and/or anxiety disorders resulted in hyperkinetic cardiovascular autonomic regulation, often associated with increased coronary risk.

DETAILED DESCRIPTION:
BACKGROUND:

Prospective epidemiologic data indicate a strong relationship of chronic anxiety and/or anxiety disorders to risk of sudden cardiac death. Other studies have shown that cardiac autonomic mechanisms are altered among stably anxious individuals in the direction of reduced parasympathetic and elevated sympathetic control. The latter investigations, however, have been based on very small clinic samples and have been incomplete in their assessment of cardiovascular regulation in anxiety.

This investigation was the first large-scale population-based research examining the cardiovascular physiology of anxiety, and helped to increase understanding of the reported association between anxiety and sudden cardiac death. This study also helped to identify groups in the general population at increased risk of sudden death.

DESIGN NARRATIVE:

The study used an ongoing well-characterized cohort, the VA Normative Aging Study (NAS), to recruit middle-aged and older community-dwelling men and women into the study. Using a variety of validated psychological and psychiatric screening instruments--including the Brief Symptom Inventory, the Composite International Diagnostic Interview, the Spielberger State-Trait Anxiety Inventory, and the Crown-Crisp Index--the study population was characterized in terms of symptoms of anxiety and diagnosis of anxiety disorders. Cardiovascular autonomic control was then assessed among anxious and non-anxious individuals using non-invasive time-domain and power-spectral measures of heart rate and blood pressure variability. Cardiac output, total peripheral resistance, and end-tidal pCO2 were simultaneously assessed.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sparrow — Brigham and Women's Hospital

REFERENCES:
- [Background] Kubzansky LD, Kawachi I, Sparrow D. Socioeconomic status, hostility, and risk factor clustering in the Normative Aging Study: any help from the concept of allostatic load? Ann Behav Med. 1999 Fall;21(4):330-8. doi: 10.1007/BF02895966. PMID 10721441
- [Background] Kubzansky LD, Kawachi I, Weiss ST, Sparrow D. Anxiety and coronary heart disease: a synthesis of epidemiological, psychological, and experimental evidence. Ann Behav Med. 1998 Spring;20(2):47-58. doi: 10.1007/BF02884448. PMID 9989308
- [Background] Siegman AW, Kubzansky LD, Kawachi I, Boyle S, Vokonas PS, Sparrow D. A prospective study of dominance and coronary heart disease in the Normative Aging Study. Am J Cardiol. 2000 Jul 15;86(2):145-9. doi: 10.1016/s0002-9149(00)00850-x. PMID 10913473